CLINICAL TRIAL: NCT01668186
Title: Longitudinal Natural History Study of Patients With Peroxisome Biogenesis Disorders (PBD)
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nancy Braverman, MD, M.Sc. Professor, Depts. of Human Genetics and Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 11-090-PED
Record Dates: First submitted 2012-08-10; First posted 2012-08-17 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Peroxisome Biogenesis Disorder; Zellweger Spectrum Disorder; RCDP - Rhizomelic Chondrodysplasia Punctata; D-Bifunctional Protein Deficiency; Alpha-Methylacyl-CoA Racemase Deficiency; Peroxisomal Acyl-CoA Oxidase Deficiency; Peroxisomal Acyl-CoA Oxidase 2 Deficiency; ATP Binding Cassette Subfamily D Member 3 Gene Mutation; ACBD5 (AcylCoA Binding Domain 5) Deficiency; Adult Refsum Disease; Sterol Carrier Protein 2 Deficiency
Keywords: Peroxisome biogenesis disorders; PBD; Zellweger spectrum disorder; Rhizomelic chondrodysplasia punctata; DBP; ACOX1; AMACR; ARD; ACBD5; ZSD; RCDP; ACOX2; ABCD3; Adult Refsum; PHYH; SCPx; RCDP1; RCDP2; RCDP3
MeSH Terms: conditions — Zellweger Syndrome; Chondrodysplasia Punctata, Rhizomelic; Pseudo-Zellweger syndrome; Alpha-Methylacyl-CoA Racemase Deficiency; Peroxisomal ACYL-COA oxidase deficiency; Refsum Disease; Peroxisome biogenesis disorders; Rhizomelic chondrodysplasia punctata, type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood, dried blood spots, urine, and specimens obtained for other e.g. cultured fibroblasts, liver biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with a peroxisomal disorder: Collection of medical records and images (ultrasounds, X-rays, MRIs, CT scans, ophthalmic images), Next-generation panel, Drug screening, and Consultation

SUMMARY:
The Peroxisome Biogenesis Disorders (PBD) are a group of inherited disorders due to defects in peroxisome assembly causing complex developmental and metabolic sequelae. In spite of advancements in peroxisome biology, the pathophysiology remains unknown, the spectrum of phenotypes poorly characterized and the natural history not yet systematically reported. Our aims are to further define this population clinically, biochemically and genetically. The investigators will prospectively follow patients from Canada, the US and internationally, and collect data from medical evaluations, blood, urine and imaging studies that would be performed on a clinical care basis. For patients who are unable to attend our clinic, we will collect all medical records and images since birth as well as subsequent records/images for the next 5 years or until the end of the study. Clinical data from medical records will be banked in our Peroxisomal Disorder Research Databank and Biobank. The investigators will use this information to identify standards of care and improve management.

DETAILED DESCRIPTION:
Participants have the option to be seen in consultation at the McGill University Health Centre in Montreal, Canada, on a yearly basis. This includes a consultation in Genetics, Nutrition, Neurology, and Ophthalmology (OCT and FAF exams). All medical records and images will be collected, retrospectively and prospectively, until the end of the study, and entered anonymously in a database. Biospecimens will be collected to identify new biomarkers. Candidate drugs will be evaluated for recovery of peroxisome functions in cultured fibroblasts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PBD or
* Single peroxisome enzyme/protein defect with phenotype similar to PBD

Exclusion Criteria:

* Not a PBD
* Not a single peroxisome enzyme/protein defect with phenotype similar to PBD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with a PBD diagnosis- or related single enzyme/protein defect
Sampling Method: Non-Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Documentation of the clinical findings | Yearly up to 10 years
  Clinical findings include but are not limited to: life span, growth parameters, development, vision, hearing, neurological examinations, renal problems, adrenal function, skeletal problems, and any other system involvement.

SECONDARY OUTCOMES:
Peroxisome function testing | Yearly up to 10 years
  To include very long chain saturated, branched and polyunsaturated fatty acids, bile acids, plasmalogens, pipecolic acid, adrenal functions, liver functions, and urine oxalate.
Development of leukodystrophy | Yearly up to 10 years
  Identification of patterns and course by MRI
Scoring of fundus photography (OCT and FAF) | Yearly up to 10 years
  Identification of patterns and course
Genotype-phenotype correlation | Yearly up to 10 years
  Correlation of mutation type to peroxisome biochemistry, number and type of disease complications.
Frequency of various disease complications and identification of risk factors in the PBD population | Yearly up to 10 years
  Neurological, vision, hearing, liver dysfunction, adrenal insufficiency, osteopenia, renal stones
Development of care management guideline resource for adolescents and adults with PBD-ZSD | Yearly up to 10 years
  Medical issues (Neurological, vision, hearing, liver dysfunction, adrenal insufficiency, osteopenia, renal stones), main challenges, and the pediatric-to-adult transition experience will be included in PBD-ZSD adult-specific management guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Braverman, MD, MS, Principal Investigator — McGill University Health Center, Montreal Childrens Hopital
Locations (1):
- Research Institute of the McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Background] Steinberg SJ, Raymond GV, Braverman NE, Moser AB. Zellweger Spectrum Disorder. 2003 Dec 12 [updated 2020 Oct 29]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1448/ PMID 20301621
- [Background] Braverman NE, Raymond GV, Rizzo WB, Moser AB, Wilkinson ME, Stone EM, Steinberg SJ, Wangler MF, Rush ET, Hacia JG, Bose M. Peroxisome biogenesis disorders in the Zellweger spectrum: An overview of current diagnosis, clinical manifestations, and treatment guidelines. Mol Genet Metab. 2016 Mar;117(3):313-21. doi: 10.1016/j.ymgme.2015.12.009. Epub 2015 Dec 23. PMID 26750748
- [Background] Braverman NE, Carroll R, Muss C, Fallatah W, Jain M. PEX7-Related Rhizomelic Chondrodysplasia Punctata. 2001 Nov 16 [updated 2025 Aug 7]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1270/ PMID 20301447
- [Background] Rush ET, Goodwin JL, Braverman NE, Rizzo WB. Low bone mineral density is a common feature of Zellweger spectrum disorders. Mol Genet Metab. 2016 Jan;117(1):33-7. doi: 10.1016/j.ymgme.2015.11.009. Epub 2015 Nov 24. PMID 26643206
- [Background] Wangler MF, Hubert L, Donti TR, Ventura MJ, Miller MJ, Braverman N, Gawron K, Bose M, Moser AB, Jones RO, Rizzo WB, Sutton VR, Sun Q, Kennedy AD, Elsea SH. A metabolomic map of Zellweger spectrum disorders reveals novel disease biomarkers. Genet Med. 2018 Oct;20(10):1274-1283. doi: 10.1038/gim.2017.262. Epub 2018 Feb 8. PMID 29419819
- [Derived] Yergeau C, Coussa RG, Antaki F, Argyriou C, Koenekoop RK, Braverman NE. Zellweger Spectrum Disorder: Ophthalmic Findings from a New Natural History Study Cohort and Scoping Literature Review. Ophthalmology. 2023 Dec;130(12):1313-1326. doi: 10.1016/j.ophtha.2023.07.026. Epub 2023 Aug 2. PMID 37541626
- [Derived] Cheung A, Argyriou C, Yergeau C, D'Souza Y, Riou E, Levesque S, Raymond G, Daba M, Rtskhiladze I, Tkemaladze T, Adang L, La Piana R, Bernard G, Braverman N. Clinical, neuroradiological, and molecular characterization of patients with atypical Zellweger spectrum disorder caused by PEX16 mutations: a case series. Neurogenetics. 2022 Apr;23(2):115-127. doi: 10.1007/s10048-022-00684-7. Epub 2022 Feb 2. PMID 35106698
- [Derived] Lee J, Yergeau C, Kawai K, Braverman N, Geleoc GSG. A Retrospective Study of Hearing Loss in Patients Diagnosed with Peroxisome Biogenesis Disorders in the Zellweger Spectrum. Ear Hear. 2022 Mar/Apr;43(2):582-591. doi: 10.1097/AUD.0000000000001126. PMID 34534157